CLINICAL TRIAL: NCT01951612
Title: Cognitive Changes and Rehabilitation in People With Transient Ischemic Attack, Stroke, or Stroke Risk Factors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baycrest (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Brian Levine, Senior Scientist, Baycrest
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08-53; 232-2009 (Other: Sunnybrook Health Sciences Centre)
Record Dates: First submitted 2013-09-24; First posted 2013-09-26 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Ischemic White Matter Disease; Transient Ischemic Attack; Mild Stroke; Stroke Risk
Keywords: cognitive impairment; ischemic white matter disease; small vessel disease; transient ischemic attack; mild stroke; stroke risk
MeSH Terms: conditions — Ischemic Attack, Transient; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Executive Function Training Program (Experimental): Participants in this group will receive the novel intervention training.
  Interventions: Behavioral: Executive Function Training Program
- Psychoeducational Training Program (Active Comparator): Participants in this group will receive the control intervention training.
  Interventions: Behavioral: Psychoeducational Training Program

INTERVENTIONS:
Behavioral: Executive Function Training Program — Participants will take part in ten 2-hour sessions over 5 weeks.
  Arms: Executive Function Training Program
Behavioral: Psychoeducational Training Program — Participants will take part in ten 2-hour sessions over 5 weeks.
  Arms: Psychoeducational Training Program

SUMMARY:
Stroke is a leading cause of disability; most strokes (80%) are subcortical, with ischemic damage due to occlusion in penetrating arteries. Although ischemic white matter disease (iWMD) may lack gross clinical manifestation, it causes significant cognitive impairment, particularly on measures of executive function, attention, and memory. This impairment is attributable to diffuse damage affecting network connections.

While there are many studies concerning rehabilitation of motor function and language in patients with large focal strokes, few studies have addressed attentional and executive functions. To our knowledge, there are no such studies on iWMD. In this study, patients will be randomized to a novel intervention for improving executive function and a control condition matched for therapist exposure. Patients will be assessed pre-intervention, post-intervention, and at long-term follow-up using a battery of behavioural and neuroimaging tasks. We predict that the novel intervention will be associated with improved executive function, as assessed behaviourally, and improved frontal network function, as assessed through neuroimaging markers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic white matter disease or small vessel disease, who have experienced a transient ischemic attack, mild stroke, or are at risk of stroke
* Fluent in English
* Able to provide informed consent to all procedures
* Sufficient motor and sensory functioning to complete all study components (with correction or assistance as required)

Exclusion Criteria:

* Substance abuse
* Other psychiatric condition (other than mood, personality, or behaviour change following onset/diagnosis of white matter disease or related condition mentioned above)
* Other medical condition suspected to influence cognition

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-11; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in neuropsychological test performance at post-intervention | Baseline and post-intervention at 10 weeks
  Performance will be assessed using standardized neuropsychological tests of processing speed, attention, executive functions, visuospatial abilities, and learning and memory. A composite measure of executive functioning derived from principal components analysis will be used as the primary outcome measure.
Change from baseline in neuropsychological test performance at 2 month follow-up | Baseline and follow-up at 2 months
  Performance will be assessed using standardized neuropsychological tests of processing speed, attention, executive functions, visuospatial abilities, and learning and memory. A composite measure of executive functioning derived from principal components analysis will be used as the primary outcome measure.

SECONDARY OUTCOMES:
Change from baseline in neuroimaging (fMRI/EEG) markers at post-intervention | Baseline and post-intervention at 10 weeks
  Measurement of fMRI and EEG signal changes at post-intervention (10 weeks) will be used. Measures of brain activation and network function will be used as secondary outcome measures.
Change from baseline in neuroimaging (fMRI/EEG) markers at 2 month follow-up | Baseline and follow-up at 2 months
  Measurement of fMRI and EEG signal changes at follow-up (2 months) will be used. Measures of brain activation and network function will be used as secondary outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Levine, PhD, Principal Investigator — Rotman Research Institute, Baycrest; Gary Turner, PhD, Principal Investigator — Sunnybrook Health Sciences Centre; Sandra Black, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Baycrest, Toronto, Ontario, Canada